CLINICAL TRIAL: NCT00769691
Title: Cerebral Autoregulation Monitoring in Adults Undergoing Cardiac Surgery: Comparison of Near Infrared Spectroscopy With Transcranial Doppler
Brief Title: Monitoring of Cerebral Blood Flow Autoregulation Using Near Infrared Spectroscopy
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HL 00012384; R01HL092259 (NIH)
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cardiacsurgery
Keywords: Cardiac surgery; Cerebral blood flow autoregulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A: Adult patients undergoing cardiac surgery

SUMMARY:
Blood flow to the brain is normally regulated to ensure a constant supply of blood with oxygen and nutrients. During heart surgery using cardiopulmonary bypass, blood pressure is kept at a level that may or may not be below an individual's lower level of brain blood flow autoregulation. If lower, the brain may be exposed to an inadequate blood flow that could result in brain damage. The purpose of this study is to examine whether monitoring with a non-invasive FDA approved device that measures oxygen saturation of the superficial layers of the brain (near infrared spectroscopy) can, when combined with blood pressure measurements, provide information on the blood pressure level where brain blood flow is not autoregulated. The goal of this research is to develop a method to individualize blood pressure during surgery to a level that is within a patient's brain blood flow autoregulation range as a means for improving outcomes for patient undergoing heart surgery.

DETAILED DESCRIPTION:
Cerebral blood flow (CBF) is normally autoregulated within a range of blood pressures, thus, allowing for a constant cerebral O2 supply commensurate with metabolic demands. The lower limit of blood pressure during general anesthesia deemed tolerable is usually empirically chosen without regard to an individual's lower autoregulatory threshold. This practice may lead to cerebral hypoperfusion in some patients placing them at risk for cerebral ischemic injury. This is particularly true during cardiac surgery using cardiopulmonary bypass where mean blood pressure is maintained at some level greater than 50 mm Hg or even lower during surgical mandated situations. This practice is concern for the rising number of aged surgical patients with cerebral vascular disease whom are prone to cerebral hypoperfusion. Individualizing blood pressure to be within the patient's autoregulatory range would more likely ensure adequate CBF during surgery. In this study we will evaluate whether real-time monitoring using a near infra-red spectroscopy (NIRS) based method accurately detects the lower CBF autoregulation threshold in patients compared with a validated, but technically more challenging method of CBF autoregulation measurement using transcranial Doppler. This approach involves continuous calculation of a moving linear regression correlation coefficient between blood pressure and cerebral O2 saturation measured with NIRS as a surrogate for CBF. A correlation coefficient, termed cerebral oximetery index, is generated and displayed versus blood pressure. When CBF is dysregulated, this correlation coefficient becomes markedly positive indicating CBF is pressure passive. We will further assess the added value of this type of monitoring to detect the lower CBF autoregulatory threshold compared with predictions based on preoperative blood pressure. These aims will be addressed in the study of 178 patients greater than 60 years of age undergoing coronary artery bypass graft surgery and/or valve surgery using cardiopulmonary bypass. Due to the many hemodynamic fluctuations during cardiac surgery, autoregulatory thresholds can be determined without administration of vasoactive drugs. Neurological complications are an important source of patient morbidity, mortality, hospital costs, and impaired quality of life after cardiac and other types of surgery. NIRS monitoring is non-invasive, continuous, requires little caregiver intervention and, thus, would have wide applicability for providing information about CBF autoregulation in a variety of clinical settings including cardiac surgery. This adoption could be enhanced with the likely development of "plug-and-play" monitors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Concordance with Doppler measure | at complesion

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Hogue, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Hori D, Katz NM, Fine DM, Ono M, Barodka VM, Lester LC, Yenokyan G, Hogue CW. Defining oliguria during cardiopulmonary bypass and its relationship with cardiac surgery-associated acute kidney injury. Br J Anaesth. 2016 Dec;117(6):733-740. doi: 10.1093/bja/aew340. PMID 27956671
- [Derived] Hori D, Brown C, Ono M, Rappold T, Sieber F, Gottschalk A, Neufeld KJ, Gottesman R, Adachi H, Hogue CW. Arterial pressure above the upper cerebral autoregulation limit during cardiopulmonary bypass is associated with postoperative delirium. Br J Anaesth. 2014 Dec;113(6):1009-17. doi: 10.1093/bja/aeu319. Epub 2014 Sep 25. PMID 25256545
- [Derived] Ono M, Zheng Y, Joshi B, Sigl JC, Hogue CW. Validation of a stand-alone near-infrared spectroscopy system for monitoring cerebral autoregulation during cardiac surgery. Anesth Analg. 2013 Jan;116(1):198-204. doi: 10.1213/ANE.0b013e318271fb10. Epub 2012 Dec 7. PMID 23223100
- [Derived] Ono M, Joshi B, Brady K, Easley RB, Zheng Y, Brown C, Baumgartner W, Hogue CW. Risks for impaired cerebral autoregulation during cardiopulmonary bypass and postoperative stroke. Br J Anaesth. 2012 Sep;109(3):391-8. doi: 10.1093/bja/aes148. Epub 2012 Jun 1. PMID 22661748
- [Derived] Brady K, Joshi B, Zweifel C, Smielewski P, Czosnyka M, Easley RB, Hogue CW Jr. Real-time continuous monitoring of cerebral blood flow autoregulation using near-infrared spectroscopy in patients undergoing cardiopulmonary bypass. Stroke. 2010 Sep;41(9):1951-6. doi: 10.1161/STROKEAHA.109.575159. Epub 2010 Jul 22. PMID 20651274